CLINICAL TRIAL: NCT01389752
Title: Effect of Activated Charcoal on the Pharmacokinetics of LY2216684 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Activated Charcoal on the Absorption of LY2216684 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12612; H9P-EW-LNCU (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2216684 without Charcoal, then with Charcoal (Experimental): Period 1: Single 18-mg (milligram) (two 9-mg tablets) oral dose of LY2216684 administered without Activated Charcoal. Period 2: Single 18-mg (two 9-mg tablets) oral dose of LY2216684 administered with single oral dose of 1 g/kg (gram/kilogram) of Activated Charcoal. Periods will be separated by a minimum of 7 days.
  Interventions: Drug: LY2216684; Drug: Activated Charcoal
- LY2216684 with Charcoal, then without Charcoal (Experimental): Period 1: Single 18-mg (two 9-mg tablets) oral dose of LY2216684 administered with single oral dose of 1 g/kg of Activated Charcoal. Period 2: Single 18-mg (two 9-mg tablets) oral dose of LY2216684 administered without Activated Charcoal. Periods will be separated by a minimum of 7 days.
  Interventions: Drug: LY2216684; Drug: Activated Charcoal

INTERVENTIONS:
Drug: LY2216684 — Administered orally
Drug: Activated Charcoal — Administered orally

SUMMARY:
The study involves a single oral dose of 18 mg (2 x 9mg tablets) LY2216684 taken on 2 occasions, once with activated charcoal and once without activated charcoal.

The study will evaluate the effect of charcoal on the absorption of LY2216684. Side effects will be documented. There will be 2 study periods each lasting up to 5 days. There will be at least 7 days between the two doses and a follow up will occur at least 7 days after the last dose. Screening is required within 30 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy, as determined by medical history and physical examination

  - Male subjects: Agree to use a reliable method of birth control during the study and for 1 month following the last dose of the study drug

  - Female subjects: Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug; or women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause (at least 1 year without menses or 6 months without menses and a follicle stimulating hormone [FSH] >40 mIU/mL [milli-international-units/milliliter])
* Have a body weight >50 kg
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling as per the protocol
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the site
* Have normal blood pressure (BP) and pulse rate (sitting position)

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product other than the investigational product used in this study; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2216684, related compounds, or any components of the formulation
* Are persons who have previously received the investigational product in this study, have completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to Screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a history or show evidence of significant active neuropsychiatric disease or have a history of suicide attempt or ideation
* Have a documented or suspected history of glaucoma
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women who are lactating
* Intend to use over-the-counter or prescription medication within 14 days prior to dosing unless deemed acceptable by the investigator and Sponsor's medical monitor. Exceptions include influenza vaccinations, the use of topical medication (provided there is no evidence of chronic dosing with the risk of systemic exposure), occasional use of acetaminophen/paracetamol/ibuprofen, hormone replacement therapy including thyroid replacement (stable dose for at least 1 month), and stable doses (at least 1 month) of oral contraceptive therapy
* Have donated blood of more than 500 mL (milliliter) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (males) or 14 units per week (females), or are unwilling to stop alcohol consumption from 48 hours prior to dosing in each period until discharge in each period (1 unit = 12 oz [ounces] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Consume 5 or more cups of coffee (or other beverages or foods of comparable caffeine content) per day, on a habitual basis, or are unwilling to stop caffeine consumption from 48 hours prior to dosing in each period until discharge in each period
* Subjects unwilling to adhere to the smoking restrictions of the Clinical Research Unit (CRU) while a resident of the CRU.
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment or are unwilling to avoid them during the study
* Subjects determined to be unsuitable by the investigator for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Study Period 1
Arm/Group | LY2216684 Without Charcoal, Then With Charcoal | LY2216684 With Charcoal, Then Without Charcoal
Started | 11 | 11
Completed | 11 | 9
Not Completed | 0 | 2
Not completed — Sponsor decision | 0 | 2
Period: Study Period 2
Arm/Group | LY2216684 Without Charcoal, Then With Charcoal | LY2216684 With Charcoal, Then Without Charcoal
Started | 11 | 9
Completed | 10 | 9
Not Completed | 1 | 0
Not completed — Sponsor decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: During Study Period 1, participants received a single oral dose of 18 mg LY2216684 alone or in combination with 1 g/kg Activated Charcoal 1 hour after LY2216684 administration. After at least 7 days, participants who initially received 18 mg LY2216684 alone received another single oral dose of 18 mg LY2216684 in combination with 1 g/kg Activated Charcoal 1 hour after LY2216684 administration during Study Period 2; participants who initially received 18 mg LY2216684 in combination with 1 g/kg Activated Charcoal received another single oral dose of 18 mg LY2216684 alone during Study Period 2.
Arm/Group | Overall
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-∞) of LY2216684
Description: The AUC0-∞ of LY2216684 was measured. The AUC was calculated for LY2216684 administered alone (reference) and LY2216684 co-administered with charcoal (test). Geometric Least Squares (LS) means were calculated according to the following model: Log(PK) = sequence + period + treatment + subject + random error for AUC.
Time Frame: Predose, up to 72 hours after administration of study drug
Population: All participants who were randomized, for whom AUC0-∞ data were available, and who were not excluded due to vomiting within twice the median time to maximum plasma concentration (tmax) of LY2216684.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nanogram*hour/milliliter (ng*h/mL)
Groups:
- LY2216684 in Combination With Activated Charcoal: Participants received a single oral dose of 18 mg (milligram) LY2216684 and a single oral dose of 1 g/kg (gram/kilogram) of Activated Charcoal 1 hour after administration of LY2216684.
- LY2216684 Alone: Participants received a single oral dose of 18 mg LY2216684.
Arm/Group | LY2216684 in Combination With Activated Charcoal | LY2216684 Alone
Number analyzed (Participants) | 17 | 19
nanogram*hour/milliliter (ng*h/mL) | 509 [454 to 571] | 786 [701 to 881]
Statistical Analysis 1: Comparison: LY2216684 in Combination With Activated Charcoal vs LY2216684 Alone; Test type: Superiority or Other; Mixed Models Analysis — The outcome was measured as a ratio of geometric means between the two treatments (LY2216684 in combination with activated charcoal/LY2216684 alone), and the 90% Confidence Interval for the ratio; Ratio of Geometric Least Squares Means = 0.65, 90% CI 2-sided [0.61 to 0.68]

2. Primary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of LY2216684
Description: The Cmax of LY2216684 was assessed. The Cmax was calculated for LY2216684 administered alone (reference) and LY2216684 co-administered with charcoal (test). Geometric LSMeans were calculated according to the following model: Log(PK) = sequence + period + treatment + subject + random error for Cmax.
Time Frame: Predose, up to 72 hours after administration of study drug
Population: All participants who were randomized, for whom Cmax data were available, and who were not excluded due to vomiting within twice the median time to maximum plasma concentration (tmax) of LY2216684.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nanogram/milliliter (ng/mL)
Groups:
- LY2216684 in Combination With Activated Charcoal: Participants received a single oral dose of 18 mg LY2216684 and a single oral dose of 1 g/kg of Activated Charcoal 1 hour after administration of LY2216684.
Arm/Group | LY2216684 in Combination With Activated Charcoal | LY2216684 Alone
Number analyzed (Participants) | 17 | 19
nanogram/milliliter (ng/mL) | 54.06 [49.16 to 59.44] | 59.84 [54.55 to 65.63]
Statistical Analysis 1: Comparison: LY2216684 in Combination With Activated Charcoal vs LY2216684 Alone; Test type: Superiority or Other; Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio of Geometric Least Squares Means = 0.90, 90% CI 2-sided [0.83 to 0.98]

3. Primary Outcome: Pharmacokinetics: Time to Maximum Plasma Concentration (Tmax) of LY2216684
Description: The tmax for LY2216684 was assessed.
Time Frame: Predose, up to 72 hours after administration of study drug
Population: All participants who were randomized, for whom tmax data were available, and who were not excluded due to vomiting within twice the median tmax of LY2216684.
Measure: Median (Full Range); unit: hours
Arm/Group | LY2216684 in Combination With Activated Charcoal | LY2216684 Alone
Number analyzed (Participants) | 17 | 17
hours | 2.00 [0.92 to 3.00] | 2.03 [2.00 to 5.00]
Statistical Analysis 1: Comparison: LY2216684 in Combination With Activated Charcoal vs LY2216684 Alone; Test type: Superiority or Other; p = 0.0010, Wilcoxon (Mann-Whitney) — The outcome was measured using the median of paired differences between the 2 treatment groups: LY2216684 administered alone (reference) versus LY2216684 co-administered with charcoal (test); Median Difference (Final Values) = -0.55, 90% CI 2-sided [-1.04 to -0.50]

ADVERSE EVENTS:
Arm/Group | LY2216684 in Combination With Activated Charcoal | LY2216684 Alone
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 9/22 | 7/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 in Combination With Activated Charcoal (N=22) | LY2216684 Alone (N=20)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/11 (1) | 1/10 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days